CLINICAL TRIAL: NCT03142776
Title: Evaluation of the Local Effect of Nonsurgical Periodontal Treatment of Generalized Aggressive Periodontitis Associated or Not With Systemic Antibiotics and Photodynamic Therapy.: a Randomized Clinical Trial
Brief Title: Nonsurgical Periodontal Treatment Associated or Not With Systemic Antibiotics and Photodynamic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, PhD, Adjunct professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLMPDT
Record Dates: First submitted 2017-05-02; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Aggressive Periodontitis, Generalized
Keywords: clarithromycin; photodynamic therapy; Antimicrobial therapy; Periodontal pocket
MeSH Terms: conditions — Aggressive Periodontitis; Periodontal Pocket | interventions — Periodontal Debridement; Photochemotherapy; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Periodontal debridement (Placebo Comparator): Periodontal pockets that received periodontal debridement associated with placebo (members took with placebo 500 mg b.i.d. for 3 days).
  Interventions: Procedure: periodontal debridement
- Periodontal debridement + CLM (Active Comparator): Periodontal pockets that received periodontal debridement associated with systemic clarithromycin (500 mg - 12/12 hours) for 3 days.
  Interventions: Procedure: periodontal debridement; Drug: systemic clarithromycin
- Periodontal debridement + PDT (Active Comparator): Periodontal pockets that received periodontal debridement associated with placebo (members took with placebo 500 mg b.i.d. for 3 days) and a single application of PDT (Photodynamic Therapy).
  Interventions: Procedure: periodontal debridement; Procedure: photodynamic therapy
- Periodontal debridement + CLM + PDT (Active Comparator): Periodontal pockets that received periodontal debridement associated with systemic clarithromycin (500 mg - 12/12 hours for 3 days) and single application of PDT.
  Interventions: Procedure: periodontal debridement; Procedure: photodynamic therapy; Drug: systemic clarithromycin

INTERVENTIONS:
Procedure: periodontal debridement
  Other Names: Ultrassonic periodontal debridement
Procedure: photodynamic therapy
  Other Names: antimicrobial photodynamic therapy
  Arms: Periodontal debridement + CLM + PDT; Periodontal debridement + PDT
Drug: systemic clarithromycin
  Other Names: antibiotic
  Arms: Periodontal debridement + CLM; Periodontal debridement + CLM + PDT

SUMMARY:
To assess the local effect of the antimicrobial therapy using clarithromycin association with photodynamic therapy (PDT) in the treatment of generalized aggressive periodontitis (GAgP).

DETAILED DESCRIPTION:
The aim of the present study was to evaluate the local effect of the antimicrobial therapy using clarithromycin (CLM) association with photodynamic therapy (PDT) in the treatment of generalized aggressive periodontitis (GAgP). Sixty periodontal pockets were select and randomly assigned into four groups: Periodontal Debridement (PD) (n=15): periodontal pockets that received periodontal debridement (PD) with placebo; PD+CLM (n=15): periodontal pockets that received periodontal debridement associated with clarithromycin; PD+PDT (n=15): periodontal pockets that received periodontal debridement associated with photodynamic therapy; PD+CLM+PDT (n=15): periodontal pockets that received periodontal debridement associated with clarithromycin and photodynamic therapy. Probing depth (PD),gain in clinical attachment level (CAL) and bleeding on probing (BOP) were evaluated at baseline, 3 and 6 months post- operatively.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of GagP
* presence of ≥20 teeth
* <35 years of age
* periodontal pockets with probing depth (PD) and Clinical Attachment Level (CAL) ≥ 5mm with concomitant bleeding on probing (BOP) in single-rooted teeth from different quadrants - agree to participate in the study and sign a written consent.

Exclusion Criteria:

* pregnant or lactating
* suffering from any other systemic disease (e.g. cardiovascular, diabetes, blood dyscrasias, immunodeficiency, etc) which could alter the course of periodontal disease
* received antimicrobials in the previous 6 months
* taking long-term anti-inflammatory drugs
* received a course of periodontal treatment within the last 12 months
* smoked

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level | 6 months
  distance from bottom of pocket to the cement-enamel junction

SECONDARY OUTCOMES:
Probing depth | 6 months
  distance from the bottom of sulcus/pocket to gingival margin

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, DDS, PhD, Study Director — UPECLIN HC FM Botucatu Unesp

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arweiler NB, Pietruska M, Pietruski J, Skurska A, Dolinska E, Heumann C, Auschill TM, Sculean A. Six-month results following treatment of aggressive periodontitis with antimicrobial photodynamic therapy or amoxicillin and metronidazole. Clin Oral Investig. 2014 Dec;18(9):2129-35. doi: 10.1007/s00784-014-1193-6. Epub 2014 Feb 4. PMID 24493231